CLINICAL TRIAL: NCT01755104
Title: A Randomized Double-blind Placebo Controlled Trial on the Effect of Stablor™ on the Abdominal Visceral Fat Mass Loss in Patients With a Metabolic Syndrome
Brief Title: Effect of Stablor on Visceral Fat Loss in Patients With a Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Nutrition et Cardiometabolisme (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCM-EFF-1
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stablor (Experimental): dietary supplement Stablor
  Interventions: Dietary Supplement: Stablor
- Placebo (Placebo Comparator): dietary supplement Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Stablor
  Arms: Stablor
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the impact of the intake of a dietary supplement STABLOR™ on the change of the abdominal visceral fat mass in patients with a metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* With a Body Mass Index (BMI) more than or equal to 25 kg/m² and less than 40 kg/m²,
* With a metabolic syndrome characterized by a a waist circumference of more than 94 cm for the males (90 cm for South-Asians, Chinese and Japanese) and more than 80 cm for the females, and at least 2 of the following criteria :

  * Arterial Blood pressure > or = 130 mmHg (systolic) and/or more than or equal to 85 mmHg (diastolic) or stabilized with treatment for at least 6 months,
  * Fasting glycemia > or = 1 g/L or 5.6 mmol/L or stabilized with treatment for at least 6 months and non-diabetic < 1.26 g/L,
  * Triglycerides > or = 1.5 g/L or 1.71 mmol/L or stabilized with treatment for at least 6 months,
  * HDL Cholesterol <0.40 g/L or 1.03 mmol/L (males) and <0,5 g/l or 1.29 mmol/L (females) or stabilized with treatment for at least 6 months.

Exclusion Criteria:

* Pregnant (positive pregnancy test at the selection visit or breast-feeding woman,
* Woman of childbearing potential without an efficient contraception method,

The above information is not intended to contain all considerations relevant to a patient's potential participation in the clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in visceral fat area assessed by computerized tomodensitometry | From baseline to Week 12

SECONDARY OUTCOMES:
Changes in selected cardiometabolic risk factors : anthropometric and physical measurements, biomarkers | from baseline to end of study
Quality of life, psychological and behavioral changes | From baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Karine Clement, MD, Principal Investigator — Institut CardioMetabolisme et Nutrition (ICAN)
Locations (2):
- Institut des Nutraceutiques et des Aliments Fonctionnels (INAF), Laval, Quebec, Canada
- Institut CardioMetabolisme et Nutrition (ICAN), Paris, France

REFERENCES:
- [Derived] Bel Lassen P, Belda E, Prifti E, Dao MC, Specque F, Henegar C, Rinaldi L, Wang X, Kennedy SP, Zucker JD, Calame W, Lamarche B, Claus SP, Clement K. Protein supplementation during an energy-restricted diet induces visceral fat loss and gut microbiota amino acid metabolism activation: a randomized trial. Sci Rep. 2021 Aug 2;11(1):15620. doi: 10.1038/s41598-021-94916-9. PMID 34341379